CLINICAL TRIAL: NCT05729568
Title: A Phase 2 Randomized, Open-label Study to Evaluate the Safety and Efficacy of Broadly Neutralizing Antibodies (bNAbs) GS-5423 and GS-2872 in Combination With the Capsid Inhibitor Lenacapavir as Long-Acting Treatment Dosed Every 6 Months in Virologically Suppressed Adults With HIV-1 Infection
Brief Title: A Study of Teropavimab and Zinlirvimab in Combination With Capsid Inhibitor Lenacapavir in Virologically Suppressed Adults With HIV-1 Infection
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-536-5939
Record Dates: First submitted 2023-02-06; First posted 2023-02-15 (Actual); Results first posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-06

CONDITIONS: HIV Infection
MeSH Terms: conditions — HIV Infections | interventions — lenacapavir; Antiretroviral Therapy, Highly Active

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Randomized Phase Treatment Group 1: LEN + TAB + ZAB (Experimental): Participants will receive loading dose of lenacapavir (LEN) 600 mg tablets, orally, on Day 1 and Day 2. They will receive LEN 927 mg subcutaneous (SC) injection along with teropavimab (TAB) 2550 mg intravenous (IV) infusion and zinlirvimab (ZAB) 2550 mg IV infusion on Day 1 and every 6 months (Q6M) up to Week 52 in the Randomized Phase.
  Interventions: Drug: Teropavimab; Drug: Zinlirvimab; Drug: Lenacapavir Tablet; Drug: Lenacapavir Injection
- Randomized Phase Treatment Group 3: SBR (Experimental): Participants in Stay on Baseline Regimen (SBR) group will continue their baseline oral antiretroviral therapy (ART) up to Week 52. ART included drugs like bictegravir/emtricitabine/tenofovir alafenamide, darunavir/cobicistat/emtricitabine/tenofovir alafenamide, dolutegravir/abacavir lamivudine, and rilpivirine/emtricitabine/tenofovir alafenamide, administered as per standard of care.
  Interventions: Drug: Antiretroviral Therapy
- Extension Phase: Treatment Group 1: LEN + TAB + ZAB (Experimental): At Week 52, participants in this group with HIV-1 RNA < 50 copies/mL will be given the option to participate in the study extension phase. In the study extension phase, participants will continue to receive their randomized study drugs every 26 weeks.
  Interventions: Drug: Teropavimab; Drug: Zinlirvimab; Drug: Lenacapavir Injection
- Extension Phase Treatment Group 3: SBR (Experimental): At Week 52, participants in this group with HIV-1 RNA < 50 copies/mL and in the absence of confirmed virologic rebound throughout the Randomized Phase of the study will be given the option to participate in the Extension Phase to switch from oral ART to LEN, TAB and ZAB, every 26 weeks at the dose specified for Treatment Group 1.
  Interventions: Drug: Teropavimab; Drug: Zinlirvimab; Drug: Lenacapavir Tablet; Drug: Lenacapavir Injection

INTERVENTIONS:
Drug: Teropavimab — Administered intravenously
  Other Names: GS-5423
  Arms: Extension Phase Treatment Group 3: SBR; Extension Phase: Treatment Group 1: LEN + TAB + ZAB; Randomized Phase Treatment Group 1: LEN + TAB + ZAB
Drug: Zinlirvimab — Administered intravenously
  Other Names: GS-2872
  Arms: Extension Phase Treatment Group 3: SBR; Extension Phase: Treatment Group 1: LEN + TAB + ZAB; Randomized Phase Treatment Group 1: LEN + TAB + ZAB
Drug: Lenacapavir Tablet — Administered orally
  Other Names: GS-6207
  Arms: Extension Phase Treatment Group 3: SBR; Randomized Phase Treatment Group 1: LEN + TAB + ZAB
Drug: Lenacapavir Injection — Administered subcutaneously
  Other Names: GS-6207; Sunlenca®
  Arms: Extension Phase Treatment Group 3: SBR; Extension Phase: Treatment Group 1: LEN + TAB + ZAB; Randomized Phase Treatment Group 1: LEN + TAB + ZAB
Drug: Antiretroviral Therapy — Antiretroviral therapy, administered orally may include regimens such as: bictegravir/emtricitabine/tenofovir alafenamide, darunavir/cobicistat/emtricitabine/tenofovir alafenamide, dolutegravir/abacavir lamivudine, and rilpivirine/emtricitabine/tenofovir alafenamide.
  Arms: Randomized Phase Treatment Group 3: SBR

SUMMARY:
The goal of this study is to test the effectiveness, safety, and tolerability of the combination of broadly neutralizing antibodies (bNAbs) (teropavimab (TAB; GS-5423) and zinlirvimab (ZAB; GS-2872)) with lenacapavir (LEN) in virologically suppressed adults with HIV-1 infection.

The purpose of this study is to evaluate the efficacy of switching to a regimen of LEN, TAB and ZAB, versus continuing on baseline oral antiretroviral therapy (ART) as determined by the proportion of participants with human immunodeficiency virus-1 (HIV-1) ribonucleic acid (RNA) ≥ 50 copies/mL at Week 26.

DETAILED DESCRIPTION:
Participants will be randomized in Treatment Groups 1 and 2 to receive LEN, TAB, and ZAB, with differing doses of TAB and ZAB between the 2 groups and in Treatment Group 3 to continue their baseline oral ART for 52 weeks. Eligible participants in Treatment Groups 1 through 3 will have the option of participating in the study extension phase to receive LEN, TAB and ZAB after completing study follow-up through Week 52.

Treatment Group 2 was removed prior to dosing of all groups during Protocol Amendment 2.

ELIGIBILITY:
Key Inclusion Criteria:

* On stable oral antiretroviral therapy (ART) consisting of no more than 2 drug classes (with the exception of pharmacologic boosters cobicistat or ritonavir) for ≥ 1 year prior to screening visit 2. A change in ART regimen ≥ 28 days prior to screening visit 2 for reasons other than virologic failure (VF) (eg, tolerability, simplification, drug-drug interaction profile) is allowed.
* No clinically significant documented historical resistance to the current ART regimen with the exception of isolated nucleoside reverse transcriptase inhibitor mutations including M184V or ≤ 2 thymidine analog mutations (TAMs: M41L, D67N, K70R, L210W, T215Y, and/or K219Q).
* Plasma human immunodeficiency virus-1 (HIV-1) ribonucleic acid (RNA) < 50 copies/mL at screening visit 2.
* Documented plasma HIV-1 RNA < 50 copies/mL for ≥ 12 months preceding screening visit 2 (or undetectable HIV-1 RNA level according to the local assay being used if the limit of detection is ≥ 50 copies/mL). Virologic elevations of ≥ 50 copies/mL (transient detectable viremia or "blips") prior to screening are acceptable.
* Proviral phenotypic sensitivity to both teropavimab and zinlirvimab at screening or from protocol GS-US-536-5816 within 24 months prior to screening.
* Screening clusters of differentiation 4 (CD4)+ T-cell count ≥ 200 cells/μL at screening visit 2.

Key Exclusion Criteria:

* Comorbid condition requiring ongoing immunosuppression.
* Evidence of hepatitis C virus (HCV) infection (prior infection cleared spontaneously or with treatment is acceptable)
* Evidence of current hepatitis B virus (HBV) infection regardless of HBV surface antigen status, at the screening visit 2.
* History of opportunistic infection or illness indicative of Stage 3 HIV disease.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-07-02 (Actual); Study Completion 2029-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (34):
- United States (29):
  - Ruane Clinical Research Group, Inc., Los Angeles, California
  - Mills Clinical Research, Los Angeles, California
  - UC San Diego (UCSD) AntiViral Research Center (AVRC), San Diego, California
  - Optimus Medical Group, San Francisco, California
  - University of Colorado Clinical and Translational Research Center, Aurora, Colorado
  - Yale University; School of Medicine; AIDS Program, New Haven, Connecticut
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Midland Florida Clinical Research Center, LLC, DeLand, Florida
  - Can Community Health Care, Fort Lauderdale, Florida
  - Midway Immunology and Research Center, Ft. Pierce, Florida
  - Orlando Immunology Center, Orlando, Florida
  - Triple O Research Institute, P.A., West Palm Beach, Florida
  - Emory University Hospital Midtown Infectious Disease Clinic, Atlanta, Georgia
  - Infectious Disease Specialists of Atlanta, Decatur, Georgia
  - Southhampton Healthcare, Inc, St Louis, Missouri
  - AXCES Research Group, LLC, Albuquerque, New Mexico
  - Montefiore Medical Center, The Bronx, New York
  - NC TraCS Institute - CTRC; University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Health Center, Durham, North Carolina
  - Regional Center for Infectious Disease Research, Greensboro, North Carolina
  - The Brody School of Medicine at East Carolina University, Greenville, North Carolina
  - Rosedale Health and Wellness, Huntersville, North Carolina
  - Prisma Health - Clinical Research Unit, Columbia, South Carolina
  - St Jude Children's Research Hospital, Memphis, Tennessee
  - Central Texas Clinical Research, Austin, Texas
  - AIDS Arms, Inc. DBA Prism Health North Texas, Dallas, Texas
  - AXCES Research Group, LLC, El Paso, Texas
  - The Crofoot Research Center, INC, Houston, Texas
  - Clinical Alliance for Research & Education, Infectious Diseases LLC (CARE-ID), Annandale, Virginia
- Australia (3):
  - East Sydney Doctors, Darlinghurst, New South Wales
  - Holdsworth House Medical Practice, Sydney, New South Wales
  - Alfred Hospital, Melbourne, Victoria
- Maple Leaf Research/Maple Leaf Medical Clinic, Toronto, Canada
- Clinical Research Puerto Rico, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mponponsuo K, McMahon JH, Gorgos L, Morales-Ramirez J, Workowski K, Brunetta J, Ogbuagu O, Collins SE, VanderVeen LA, Huang H, Baeten JM, Eron JJ. Efficacy and Safety of Lenacapavir, Teropavimab, and Zinlirvimab: Phase II Week 26 Primary Outcome [Oral 07]. Conference on Retroviruses and Opportunistic Infections (CROI); 2025 9-12 March, San Francisco, CA.
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=GS-US-536-5939

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 241 participants were screened. The study planned to enroll participants in Treatment Groups 1, 2 and 3. However, per review of the programmatic data overall and from study GS-US-536-5816 (NCT04811040), Treatment Group 2 was removed prior to dosing of all groups in the study and did not enroll any participants. Therefore, data is reported only for Treatment Groups 1 and 3.
Pre-assignment Details: Participants were enrolled at study sites in the United States, Puerto Rico, Australia, and Canada.
  Data submitted represent primary analysis performed on data collected by the Primary Analysis Completion Date (02-July-2024). Complete data will be submitted within 1 year of actual study completion date.
Groups:
- Randomized Phase Treatment Group 1: LEN + TAB + ZAB: Participants received loading dose of Lenacapavir (LEN) 600 mg tablets, orally, on Day 1 and Day 2. They received LEN 927 mg subcutaneous (SC) injection along with teropavimab (TAB) 2550 mg intravenous (IV) infusion and zinlirvimab (ZAB) 2550 mg IV infusion on Day 1 and every 6 months (Q6M) or every 26 weeks (Q26W) up to Week 52 in the Randomized Phase.
  At Week 52, participants in this group with HIV-1 RNA < 50 copies/mL are given the option to participate in the study extension phase. In the study extension phase, participants continued to receive their randomized study drugs every 26 weeks.
- Randomized Phase Treatment Group 3: SBR: Participants in Stay on Baseline Regimen (SBR) group continued their baseline oral antiretroviral therapy (ART) up to Week 52. Antiretroviral therapy included drugs like bictegravir/emtricitabine/tenofovir alafenamide, darunavir/cobicistat/emtricitabine/tenofovir alafenamide, dolutegravir/abacavir lamivudine, and rilpivirine/emtricitabine/tenofovir alafenamide, administered as per standard of care.
  At Week 52, participants in this group with HIV-1 RNA < 50 copies/mL and in the absence of confirmed virologic rebound throughout the Randomized Phase of the study are given the option to participate in the Extension Phase to switch from ART to LEN, TAB and ZAB, every 26 weeks at the dose specified for Treatment Group 1.
Period: Overall Study
Arm/Group | Randomized Phase Treatment Group 1: LEN + TAB + ZAB | Randomized Phase Treatment Group 3: SBR
Started | 56 | 27
Completed | 0 | 0
Not Completed | 56 | 27
Not completed — Still on Study | 52 | 26
Not completed — Randomized but Never Treated | 3 | 0
Not completed — Adverse Event | 0 | 1
Not completed — Investigator's Discretion | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all participants who were randomized and received at least 1 dose of study drug (ie, study treatment, including LEN, teropavimab, zinlirvimab, or continued with their baseline ART regimen).
Groups:
- Randomized Phase Treatment Group 1: LEN + TAB + ZAB: Participants received loading dose of LEN 600 mg tablets, orally, on Day 1 and Day 2. They received LEN 927 mg SC injection along with TAB 2550 mg IV infusion and ZAB 2550 mg IV infusion on Day 1 and Q6M up to Week 52 in the Randomized Phase.
  At Week 52, participants in this group with HIV-1 RNA < 50 copies/mL are given the option to participate in the study extension phase. In the study extension phase, participants continued to receive their randomized study drugs every 26 weeks.
- Randomized Phase Treatment Group 3: SBR: Participants in SBR group continued their baseline oral ART up to Week 52. Antiretroviral therapy included drugs like bictegravir/emtricitabine/tenofovir alafenamide, darunavir/cobicistat/emtricitabine/tenofovir alafenamide, dolutegravir/abacavir lamivudine, and rilpivirine/emtricitabine/tenofovir alafenamide, administered as per standard of care.
  At Week 52, participants in this group with HIV-1 RNA < 50 copies/mL and in the absence of confirmed virologic rebound throughout the Randomized Phase of the study are given the option to participate in the Extension Phase to switch from ART to LEN, TAB and ZAB, every 26 weeks at the dose specified for Treatment Group 1.
- Total: Total of all reporting groups
Arm/Group | Randomized Phase Treatment Group 1: LEN + TAB + ZAB | Randomized Phase Treatment Group 3: SBR | Total
Number analyzed (Participants) | 53 | 27 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 52 | 26 | 78
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (13.7) | 53 (9.6) | 47 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 12
  Male | 45 | 23 | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 7 | 20
  Not Hispanic or Latino | 40 | 20 | 60
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 21 | 8 | 29
  White | 28 | 16 | 44
  More than one race | 3 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 48 | 19 | 67
  Australia | 2 | 6 | 8
  Puerto Rico | 2 | 1 | 3
  Canada | 1 | 1 | 2
Clusters of Differentiation 4 (CD4)+ T-cell Counts [Mean (Standard Deviation); unit: cells/µL] | 740 (239.3) | 768 (260.0) | 749 (245.2)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Human Immunodeficiency Virus Type 1 (HIV-1) Ribonucleic Acid (RNA) ≥ 50 Copies/mL at Week 26 as Determined by the United States Food and Drug Administration (US FDA)-Defined Snapshot Algorithm
Description: Percentage of participants with HIV-1 RNA ≥ 50 copies/mL at Week 26 was analyzed using US FDA-defined snapshot algorithm, which defines a participant's virologic outcome and included participants a) who had last available on-treatment HIV-1 RNA ≥ 50 copies/mL in the Week 26 analysis window; b) who did not have on-treatment HIV-1 RNA data in the Week 26 analysis window and i) discontinued study drug prior to or in the Week 26 analysis window due to lack of efficacy, or ii) discontinued study drug prior to or in the Week 26 analysis window due to adverse event (AE) or death and had last available on-treatment HIV-1 RNA ≥ 50 copies/mL, or iii) discontinued study drug prior to or in the Week 26 analysis window due to reasons other than AE, death, or lack of efficacy and had the last available on-treatment HIV-1 RNA ≥ 50 copies/mL.
  Clopper-Pearson exact method was used to calculate the 95% confidence interval (CI) for the outcome measure of each treatment. Percentages were rounded off.
Time Frame: Week 26
Population: Participants in the Full Analysis Set were analyzed. The Full Analysis Set included all randomized participants who have received at least one dose of the complete long acting study drug regimen (ie, SC LEN + TAB, ZAB) or continued with their baseline ART regimen.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Randomized Phase Treatment Group 1: LEN + TAB+ ZAB: Participants received loading dose of LEN 600 mg tablets, orally, on Day 1 and Day 2. They received LEN 927 mg SC injection along with TAB 2550 mg IV infusion and ZAB 2550 mg IV infusion on Day 1 and Q6M up to Week 52 in the Randomized Phase.
  At Week 52, participants in this group with HIV-1 RNA < 50 copies/mL are given the option to participate in the study extension phase. In the study extension phase, participants continued to receive their randomized study drugs every 26 weeks.
- Randomized Phase Treatment Group 3: SBR: Participants in SBR group continued their baseline oral ART up to Week 52. Antiretroviral therapy included drugs like bictegravir/emtricitabine/tenofovir alafenamide, darunavir/cobicistat/emtricitabine/tenofovir alafenamide, dolutegravir/abacavir lamivudine, and rilpivirine/emtricitabine/tenofovir alafenamide, administered as per standard of care.
  At Week 52, participants in this group with HIV-1 RNA < 50 copies/mL and in the absence of confirmed virologic rebound throughout the Randomized Phase of the study are given the option to participate in the Extension Phase to switch from oral ART to LEN, TAB and ZAB, every 26 weeks at the dose specified for Treatment Group 1.
Arm/Group | Randomized Phase Treatment Group 1: LEN + TAB+ ZAB | Randomized Phase Treatment Group 3: SBR
Number analyzed (Participants) | 53 | 27
percentage of participants | 1.9 [0.0 to 10.1] | 0.0 [0.0 to 12.8]

2. Secondary Outcome: Percentage of Participants With HIV-1 RNA ≥ 50 Copies/mL at Week 52 as Determined by the US FDA-defined Snapshot Algorithm
Time Frame: Week 52
Reporting Status: Not Posted

3. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 26 as Determined by the US FDA-defined Snapshot Algorithm
Description: Percentage of participants with HIV-1 RNA < 50 copies/mL at Week 26 was analyzed using the US FDA-defined snapshot algorithm, which defined a participant's virologic outcome and included participants who had the last available on-treatment HIV-1 RNA < 50 copies/mL in the Week 26 analysis window.
  The Clopper-Pearson exact method was used to calculate the 95% CI for the outcome measure of each treatment. Percentages were rounded off.
Time Frame: Week 26
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Randomized Phase Treatment Group 1: LEN + TAB + ZAB | Randomized Phase Treatment Group 3: SBR
Number analyzed (Participants) | 53 | 27
percentage of participants | 96.2 [87.0 to 99.5] | 96.3 [81.0 to 99.9]

4. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 52 as Determined by the US FDA-defined Snapshot Algorithm
Time Frame: Week 52
Reporting Status: Not Posted

5. Secondary Outcome: Change From Baseline in Clusters of Differentiation 4 (CD4) + T-cell Counts at Week 26
Time Frame: Baseline, Week 26
Population: Participant in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | Randomized Phase Treatment Group 1: LEN + TAB + ZAB | Randomized Phase Treatment Group 3: SBR
Number analyzed (Participants) | 52 | 26
cells/µL | 23 (143.4) | 74 (202.6)
Statistical Analysis 1: Comparison: Randomized Phase Treatment Group 1: LEN + TAB + ZAB vs Randomized Phase Treatment Group 3: SBR; Test type: Superiority; p = 0.1436, ANCOVA; Difference in least-squares means = -56, 95% CI 2-sided [-132 to 20] — Difference in least-squares means (Diff in LSM), and its 95% CI were from ANCOVA model of change from baseline CD4 cell count with treatment as fixed effect and baseline CD4 cell count as a covariate

6. Secondary Outcome: Change From Baseline in CD4+ T-cell Counts at Week 52
Time Frame: Baseline, Week 52
Reporting Status: Not Posted

7. Secondary Outcome: Percentage of Participants Experiencing Treatment-emergent Adverse Events (TEAEs)
Time Frame: Up to approximately 6 years
Reporting Status: Not Posted

8. Secondary Outcome: Trough Concentration at Week 26 for TAB and ZAB
Description: Trough concentration is defined as the concentration of the drug in plasma/serum at the end of the dosing interval.
Time Frame: Week 26
Population: Participants in the TAB PK Analysis Set and ZAB PK Analysis Set with available data were analyzed.
  TAB PK Analysis Set included all randomized participants who have received at least 1 dose of study drug, and have at least 1 non-missing TAB concentration value reported by the PK laboratory test.
  ZAB PK Analysis Set included all randomized participants who have received at least 1 dose of study drug, and have at least 1 non-missing ZAB concentration value reported by the PK laboratory test.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Randomized Phase Treatment Group 1: LEN + TAB + ZAB
Number analyzed (Participants) | 52
µg/mL
  TAB | 41.8 (22.7)
  ZAB | 72.0 (39.2)

9. Secondary Outcome: Trough Concentration at Week 26 for LEN
Description: Trough concentration is defined as the concentration of the drug in plasma/serum at the end of the dosing interval.
Time Frame: Week 26
Population: Participants in the LEN PK Analysis Set with available data were analyzed. LEN PK Analysis Set included all randomized participants who have received at least 1 dose of study drug, and have at least 1 nonmissing LEN concentration value reported by the PK laboratory test.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Randomized Phase Treatment Group 1: LEN + TAB+ ZAB
Number analyzed (Participants) | 52
ng/mL | 20.2 (10.6)

10. Secondary Outcome: Trough Concentration at Week 52 for TAB and ZAB
Description: Trough concentration is defined as the concentration of the drug in plasma/serum at the end of the dosing interval.
Time Frame: Week 52
Reporting Status: Not Posted

11. Secondary Outcome: Trough Concentration at Week 52 for LEN
Description: Trough concentration is defined as the concentration of the drug in plasma/serum at the end of the dosing interval.
Time Frame: Week 52
Reporting Status: Not Posted

12. Secondary Outcome: Pharmacokinetic (PK) Parameter: AUC0-tau for TAB and ZAB
Description: AUC0-tau is defined as the partial area under the concentration versus time curve from time "0" to time "t".
Time Frame: Up to approximately 6 years
Reporting Status: Not Posted

13. Secondary Outcome: PK Parameter: t1/2 for TAB and ZAB
Description: t1/2 is defined as the terminal elimination half-life.
Time Frame: Up to approximately 6 years
Reporting Status: Not Posted

14. Secondary Outcome: PK Parameter: Cmax for TAB and ZAB
Description: Cmax is defined as the maximum observed concentration of drug.
Time Frame: Up to approximately 6 years
Reporting Status: Not Posted

15. Secondary Outcome: PK Parameter: Cmax for LEN
Description: Cmax is defined as the maximum observed concentration of drug.
Time Frame: Up to approximately 6 years
Reporting Status: Not Posted

16. Secondary Outcome: PK Parameter: Tmax for TAB, ZAB, and LEN
Description: Tmax is defined as the time (observed time point) of Cmax.
Time Frame: Up to approximately 6 years
Reporting Status: Not Posted

17. Secondary Outcome: Percentage of Participants With Treatment-emergent Anti-TAB and Anti-ZAB Antibodies
Description: Anti-TAB and anti-ZAB antibodies incidence referred to the percentage of participants who have treatment-emergent anti-TAB and anti-ZAB antibodies among all participants evaluable for anti-drug antibody (ADA) incidence.
Time Frame: Up to approximately 6 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: All-cause Mortality and Adverse events: Up to Week 26
Description: All-cause mortality: The All Randomized Analysis Set included all participants who were randomized into the study.
  Adverse events: The Safety Analysis Set included all participants who were randomized and received at least 1 dose of study drug (ie, study treatment, including LEN, TAB, ZAB, or continued with their baseline ART regimen).
Arm/Group | Randomized Phase Treatment Group 1: LEN + TAB + ZAB | Randomized Phase Treatment Group 3: SBR
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/53 | 1/27
Other Adverse Events (participants affected / at risk) | 40/53 | 4/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Randomized Phase Treatment Group 1: LEN + TAB + ZAB (N=53) | Randomized Phase Treatment Group 3: SBR (N=27)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Randomized Phase Treatment Group 1: LEN + TAB + ZAB (N=53) | Randomized Phase Treatment Group 3: SBR (N=27)
Constipation (Gastrointestinal disorders) | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 1
Injection site erythema (General disorders) | 11 | 0
Injection site induration (General disorders) | 7 | 0
Injection site mass (General disorders) | 3 | 0
Injection site nodule (General disorders) | 22 | 0
Injection site pain (General disorders) | 12 | 0
Covid-19 (Infections and infestations) | 1 | 2
Sinusitis (Infections and infestations) | 3 | 1
Upper respiratory tract infection (Infections and infestations) | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2024-05-13): https://cdn.clinicaltrials.gov/large-docs/68/NCT05729568/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-12): https://cdn.clinicaltrials.gov/large-docs/68/NCT05729568/SAP_001.pdf